CLINICAL TRIAL: NCT02574858
Title: Study of the Safety of QRH-882260 Heptapeptide
Acronym: QRH-882260
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00099903
Record Dates: First submitted 2015-10-07; First posted 2015-10-14 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- QRH-886620 (Experimental): The first three subjects will squirt via syringe into their mouths (po) 4.2 mg (2.1ml) mg of reconstituted (with 5 ml of 0.9% saline) QRH-882260 heptapeptide (~100 µM concentration). They will be asked to wait 5 minutes and then drink at least 4-8oz of tap water. The remaining seven subjects will receive (squirted via syringe into their mouths) 1mg (5ml) of reconstituted (with 5ml of 0.9% saline) QRH-882260 heptapeptide (~100 µM concentration).
  Interventions: Drug: QRH-882260

INTERVENTIONS:
Drug: QRH-882260 — The investigational agent to be used in this study is a fluorescently-labeled peptide composed of a 7-amino acid sequence attached to Cy5.

SUMMARY:
The purpose of this study is to evaluate the safety of orally administered QRH-882260, a topically administered Cy5-labeled heptapeptide specific for epithelial growth factor receptor (EGFR).

DETAILED DESCRIPTION:
This is a Phase IA study of the safety of an orally administered QRH-882260 heptapeptide for detection of neoplastic tissues in multiple areas of the gastrointestinal tract in humans. The investigators intend to enroll 10 evaluable subjects. The investigators expect to be able to enroll about 1-2 subjects per week, so the study should take about 1-2 months to complete.

Interested, healthy subjects ages 25-100 who respond to recruitment advertising and appear to be eligible based on a screening questionnaire will be scheduled for a study visit at MCRU. At the study visit, the subjects will review and sign the informed consent and eligibility will be confirmed. If eligible, subjects will provide a blood sample for clinical labs and a urine sample for urinalysis. A baseline EKG will be recorded. A negative urine pregnancy test for women of child-bearing potential is required to be eligible. Eligible subjects will consume the reconstituted QRH-882260 heptapeptide. After 5 minutes, subjects will drink a minimum 4-8 ounces of tap water. Subjects will remain in MCRU for observation for 30 minutes. Vital signs and an EKG will be recorded after 30 minutes. Subjects are required to have repeat blood draw for clinical labs and urinalysis within 24 to 48 hours after QRH-882260 heptapeptide ingestion. The study team will conduct a follow up phone call to verbally assess toxicity after post-ingestion labs (within 7 days).

ELIGIBILITY:
Inclusion Criteria

* Adults age 25 to 100 years
* Not pregnant (willing to have pregnancy test if applicable)
* No recent illness (infection, URI, virus or flu) within 2 weeks,
* Stable health status (i.e. no medication changes within 2 months, no recent surgery, etc. per PI)
* Willing and able to sign informed consent
* Willing and able to drink the peptide and a tap water chaser
* Willing and able to get baseline and 24-48 hours post ingestion labs Exclusion Criteria
* Known allergy to Cy5 or derivatives, such as indocyanine green (ICG)
* Subjects on active chemotherapy or radiation therapy
* Diabetics on insulin/hypoglycemic (due to fasting requirements)

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QRH-886620
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | QRH-886620
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants]
  Ages of Participants: 22-29 years | 4
  Ages of Participants: 30-39 years | 2
  Ages of Participants: 40-49 years | 5
  Ages of Participants: 50-59 years | 8
  Ages of Participants: 60-69 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Abnormal Lab Values
Description: Review of laboratory values for abnormalities after intervention with QRH-882260. If the first post-procedure labs are outside normal range, they must be within 20% of the subject's baseline lab values or returning towards normal range. Lab values not meeting these criteria must be repeated weekly until they peak and weekly until normal or within 20% of baseline level or within normal range.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- QRH-886620: The first three subjects will squirt via syringe into their mouths (po) 4.2 mg (2.1ml) mg of reconstituted (with 5 ml of 0.9% saline) QRH-882260 heptapeptide (~100 µM concentration). They will be asked to wait 5 minutes and then drink at least 4-8oz of tap water. The remaining 22 subjects will receive (squirted via syringe into their mouths) 1mg (5ml) of reconstituted (with 5ml of 0.9% saline) QRH-882260 heptapeptide (~100 µM concentration).
  QRH-882260: The investigational agent to be used in this study is a fluorescently-labeled peptide composed of a 7-amino acid sequence attached to Cy5.
Arm/Group | QRH-886620
Number analyzed (Participants) | 25
Participants | 1

2. Primary Outcome: Number of Subjects With Abnormal EKG
Description: Review of EKG for abnormalities after intervention with QRH-882260. Paired EKGs will be reviewed for electrical changes post QRH-882260 ingestion.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | QRH-886620
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Arm/Group | QRH-886620
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QRH-886620 (N=25)
Elevated creatinine level (Renal and urinary disorders) | 1 (1) — Elevated creatinine level at visit 2 of 20%. Subject returned to submit another sample for repeat testing. Creatinine level returned to within 20% of baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No